CLINICAL TRIAL: NCT01621373
Title: Prospective Exploratory Dose-finding Study in Neonates Receiving a Single Intravenous Propofol Bolus for Endotracheal Intubation During (Semi-)Elective INSURE Procedure or Non-INSURE Procedures in Neonates
Brief Title: Exploratory Propofol Dose Finding Study In Neonates
Acronym: NEOPROP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s54472; 2012-002648-26 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-18 (Estimated); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2012-08

CONDITIONS: Adverse Reaction to Drug; Neonatal Disorder
Keywords: neonatology; intratracheal intubation; propofol
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Infant, Newborn, Diseases | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- propofol (Other): All patients receive propofol. Dose will be defined based on response of previous patient in the same stratum.
  Interventions: Drug: propofol administration

INTERVENTIONS:
Drug: propofol administration — Single IV bolus propofol start at 1 mg/kg. Dose will be adapted based on predefined scoring systems with +/-0.5 mg/kg.
  Other Names: Diprivan

SUMMARY:
The aim of the study is to explore the optimal propofol dose in neonates receiving a single intravenous propofol bolus for endotracheal intubation during (semi-)elective INSURE (intubation-surfactant-extubation) procedure (preterm neonates) and (semi-)elective non-INSURE procedures (term-preterm neonates).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the pharmacokinetics and pharmacodynamics of propofol (short acting anesthetic) in 50 neonates to whom the drug is administered as a intravenous bolus. This is part of routine clinical care in patients receiving (semi-) elective intubation. It's the aim to explore the most effective IV propofol dose for a successful INSURE (intubation, surfactant, extubation) procedure and for successful (semi-) elective intubation in non-INSURE procedures. We hereby aim to define the most optimal dose regimen for propofol in neonates.

Intubation condition score was assessed retrospectively by the intubating physician.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the Neonatal Intensive Care Unit who need short procedural sedation for (semi-) elective intubation will be considered for inclusion, after informed written consent of the parents.
* Patients can be included if they are hemodynamically stable and did not receive sedative or analgesic agents during the previous 24 hours.

Exclusion Criteria:

* Known propofol intolerance

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Thewissen, MD, Principal Investigator — UZ Leuven, Belgium
Locations (1):
- Neonatal Intensive Care Unit UZ Leuven, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Smits A, Thewissen L, Caicedo A, Naulaers G, Allegaert K. Propofol Dose-Finding to Reach Optimal Effect for (Semi-)Elective Intubation in Neonates. J Pediatr. 2016 Dec;179:54-60.e9. doi: 10.1016/j.jpeds.2016.07.049. Epub 2016 Sep 2. PMID 27597733

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Propofol
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: day] | 1 [1 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Region of Enrollment [Number; unit: participants]
  Belgium | 50

OUTCOME MEASURES:

1. Primary Outcome: Effective Dose for 50% of Patients for Succesful Intubation and Subsequent Extubation in Case of Planned Extubation After INSURE Procedure
Description: An up-and-down dose-response design was used to calculate ED50 (mg/kg) in strata with effective sampling size of at least 6, by use of the Dixon-Massey method for small samples.
Time Frame: 1 hour after propofol administration
Population: Of the 8 strata defined by postmenstrual age and postnatal age, primary outcome of propofol ED 50 in mg/dl could be calculated in stratum 1,3 and 5.
Measure: Mean (95% Confidence Interval); unit: mg/kg
Groups:
- Stratum 1: Postmenstrual age < 28 w Postnatal age < 10 days
- Stratum 3: Postmenstrual age 28 to< 32 w Postnatal age < 10 days
- Stratum 5: Postmenstrual age 32 to < 37 w Postnatal age < 10 days
Arm/Group | Stratum 1 | Stratum 3 | Stratum 5
Number analyzed (Participants) | 12 | 23 | 12
mg/kg | 0.792 [0.392 to 1.192] | 0.713 [0.424 to 1.002] | 1.350 [0.932 to 1.767]

2. Other Pre Specified Outcome: Intubation Condition Score
Description: Intubation condition score at final intubation was assessed retrospectively by the intubating physician. The score as described by Viby-Mogensen was used, with the evaluation of laryngoscopy, vocal cords, coughing, jaw relaxation and limb movements. The minimum score of the intubation condition score is 5, the maximum score of the intubation condition score is 20. A score less or equal to 10 defines a good intubation condition.
Time Frame: After final intubation.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Group 1: Postmenstrual age < 28 w
- Group 2: Postmenstrual age 28 to< 32 w
- Group 3: Postmenstrual age 32 to < 37 w
- Group 4: Postmenstrual age >or = 37 w
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 12 | 24 | 12 | 2
score on a scale | 7 [5 to 13] | 6 [5 to 11] | 8 [5 to 11] | 8 [7 to 9]

ADVERSE EVENTS:
Groups:
- All Particpants: Permissive hypotension was noted with a duration of blood pressure decrease at least 120-200 minutes after propofol administration.
Arm/Group | All Particpants
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No